CLINICAL TRIAL: NCT00511225
Title: Effects of Oral Cholecalciferol (Vitamin D3) on Bone Health, Neuromuscular Function, and Quality of Life in Adults With Chronic Kidney Disease
Acronym: Neph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Principal Investigator, Laura Armas, Assistant Professor, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-14571
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: End Stage Renal Disease
Keywords: dialysis; Vitamin D
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Will receive 10,000 IU of cholecalciferol weekly
  Interventions: Dietary Supplement: cholecalciferol
- 2 (Placebo Comparator): Will receive a identical appearing placebo weekly
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol — 10,000 IU weekly
  Other Names: Maximum D3®,Pro-Pharma LLA, Kirksville, MO
  Arms: 1
Dietary Supplement: placebo — placebo capsule
  Arms: 2

SUMMARY:
Will oral vitamin improve strength, bone quality, pain and quality of life. This is a double blind, randomized placebo controlled study using 10,000 IU of cholecalciferol vs placebo.

DETAILED DESCRIPTION:
The proposed study is be a randomized, double-blind, placebo-controlled trial of supplementation with oral vitamin D3.

Each subject will take a once-weekly capsule containing vitamin D3 or a an identical-appearing placebo for a treatment period of 15 weeks.

Subjects will be assessed for Bone pain and tenderness, Neuromuscular function, physical performance score, and Quality of life assessment.

A subset of subjects will have bone biopsies performed before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* On dialysis
* Likely to be able to complete the study
* At least minimally ambulatory, with or without a walking aid (i.e., cane or walker)
* Able to complete the various questionnaires interactively with the research nurse
* Venous access that can be accomplished without unusual difficulty.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-09; Primary Completion 2010-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
change in physical performance score | 15 weeks

SECONDARY OUTCOMES:
Bone pain and tenderness | 15 weeks
Neuromuscular function tests | 15 weeks
Quality of life assessment | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lund, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Graeff-Armas LA, Kaufmann M, Lyden E, Jones G. Serum 24,25-dihydroxyvitamin D3 response to native vitamin D2 and D3 Supplementation in patients with chronic kidney disease on hemodialysis. Clin Nutr. 2018 Jun;37(3):1041-1045. doi: 10.1016/j.clnu.2017.04.020. Epub 2017 Apr 30. PMID 28506446
- [Derived] Armas LA, Andukuri R, Barger-Lux J, Heaney RP, Lund R. 25-Hydroxyvitamin D response to cholecalciferol supplementation in hemodialysis. Clin J Am Soc Nephrol. 2012 Sep;7(9):1428-34. doi: 10.2215/CJN.12761211. Epub 2012 Jul 12. PMID 22798536